CLINICAL TRIAL: NCT01138423
Title: A Randomized, Placebo-controlled, Double Blind, 4-period, Cross-over Trial, to Study the Effects of Aliskiren, Hydrochlorothiazide and Moxonidine on Endothelial Dysfunction in Obesity Related Hypertension
Brief Title: Treatment of Adiposity Related hypErTension (TARGET)
Acronym: TARGET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: dr. W. Spiering, University Medical Center Utrecht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCU-Vasc-14A
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension; Abdominal Obesity; Metabolic Syndrome
Keywords: Hypertension; Metabolic Syndrome X; Obesity; Adiposity; Clinical trial
MeSH Terms: conditions — Hypertension; Obesity, Abdominal; Metabolic Syndrome; Obesity | interventions — aliskiren; moxonidine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren; Drug: Placebo (for moxonidine and hydrochlorothiazide)
- Moxonidine (Experimental)
  Interventions: Drug: Moxonidine; Drug: Placebo (for aliskiren)
- Hydrochlorothiazide (Experimental)
  Interventions: Drug: Hydrochlorothiazide; Drug: Placebo (for aliskiren)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (for aliskiren); Drug: Placebo (for moxonidine and hydrochlorothiazide)

INTERVENTIONS:
Drug: Aliskiren — Once daily treatment with aliskiren for 8-weeks, according to the following regiment: once daily (morning time) 150 mg during the first 2 weeks, followed by once daily (morning time) 300 mg during the remaining 6 weeks. Coincidental intake of grapefruit(juice) should be avoided. This treatment interval is followed by a one-week tapering period: 150 mg on day 1, 2, 3, 4, 5 and 7.
  Other Names: Brand name: Ralisez; ATC-code: C09XA02
  Arms: Aliskiren
Drug: Moxonidine — Once daily treatment with moxonidine for 8-weeks, according to the following regiment: once daily (morning time) 0.2 mg during the first 2 weeks, followed by once daily (morning time) 0.4 mg during the remaining 6 weeks. Coincidental intake of grapefruit(juice) should be avoided. This treatment interval is followed by a one-week tapering period: 0.2 mg on day 1, 2, 3, 4, 5 and 7.
  Other Names: No brand name (generic product); ATC-code: C02AC05
  Arms: Moxonidine
Drug: Hydrochlorothiazide — Once daily treatment with hydrochlorothiazide for 8-weeks, according to the following regiment: once daily (morning time) 12.5 mg during the first 2 weeks, followed by once daily (morning time) 25 mg during the remaining 6 weeks. Coincidental intake of grapefruit(juice) should be avoided. This treatment interval is followed by a one-week tapering period: 12.5 mg on day 1, 2, 3, 4, 5 and 7.
  Other Names: No brand name (generic product); ATC-code: C03AA03
  Arms: Hydrochlorothiazide
Drug: Placebo (for aliskiren) — Once daily treatment with placebo tablets for 8-weeks, according to the following regiment: once daily (morning time) 1 tablet during the first 2 weeks, followed by once daily (morning time) 2 tablets during the remaining 6 weeks. Coincidental intake of grapefruit(juice) should be avoided. This treatment interval is followed by a one-week tapering period: 1 tablet on day 1, 2, 3, 4, 5 and 7.
  Arms: Hydrochlorothiazide; Moxonidine; Placebo
Drug: Placebo (for moxonidine and hydrochlorothiazide) — Once daily treatment with placebo capsules for 8-weeks, according to the following regiment: once daily (morning time) 1 capsule during the first 2 weeks, followed by once daily (morning time) 2 capsules during the remaining 6 weeks. Coincidental intake of grapefruit(juice) should be avoided. This treatment interval is followed by a one-week tapering period: 1 tablet on day 1, 2, 3, 4, 5 and 7.
  Arms: Aliskiren; Placebo

SUMMARY:
High blood pressure (hypertension) is an important cause of myocardial infarction and stroke. High blood pressure often occurs in people who are overweight. These people frequently also have abnormal fat and sugar metabolism. The combination of these problems is called the 'metabolic syndrome'.

People with hypertension and obesity currently receive the same drug therapy as people with hypertension, but without obesity. Different classes of drugs are thought to be equally effective in lowering blood pressure.

Next to lowering blood pressure, hypertension treatment can have additional effects, like changes in blood vessel function (the ability to dilate and constrict) or changes is the metabolism of sugar and fat. Particularly in patients with the metabolic syndrome, these additional effects are thought to be of great importance, because they can influence the risk for cardiovascular diseases.

The blood pressure lowering mechanism differs between classes of blood pressure lowering medication. The purpose of this study is to compare the effects of three types of blood pressure lowering medication belonging to different classes. The main outcomes of interest will be blood vessel function (the ability to dilate and constrict) and blood pressure. Moreover, the effect of treatment on additional outcomes, like metabolism of sugar and fat, will be studied.

DETAILED DESCRIPTION:
Treatment of obesity related hypertension (ORH) is challenging and has become an important global health problem. According to guidelines, most classes of antihypertensives are equally effective for the treatment of hypertension. However, these guidelines are based on evidence from studies in patients with essential hypertension, but without a specific focus on ORH. There is an increasing body of evidence about the complex pathophysiological mechanisms of ORH. Adipose tissue dysfunction is commonly regarded as a common soil that eventually causes up regulation of the sympathetic nervous system (SNS) and the renin-angiotensin-system (RAS). Moreover, development of hypertension is closely related to development of endothelial dysfunction, dyslipidemia and disorders of glucose metabolism. The investigators hypothesize that treatment with antihypertensives that are directed at down regulation of the SNS (moxonidine) and the RAS (aliskiren) will result in more beneficial effects than treatment with a diuretic (hydrochlorothiazide), because the latter reduces blood pressure by inhibition of sodium resorption, without influencing the underlying disease mechanism. The main outcomes of interest are endothelial function and blood pressure, but many secondary outcomes are studied too.

ELIGIBILITY:
Inclusion criteria:

* Patient is a male or post menopausal female, 30-70 years of age on the day of signing informed consent. Post menopausal status is assumed if a woman has not experienced a menstrual bleed for a minimum of 12 months, assuming that she still has a uterus, and is not pregnant or lactating. In women without a uterus, menopause or postmenopause is defined by a very high FSH level.
* All patients should fulfil the diagnostic criterion of abdominal adiposity: waist circumference > 102 cm (men) or > 88 cm (women). The waist circumference is measured halfway between the lower rib and iliac crest in standing position.
* All patients should fulfil the diagnostic criterium for hypertension: systolic blood pressure >/= 130 mmHg and/or diastolic blood pressure >/= 85 mmHg during both visits. Blood pressure is assessed by office readings in accordance with current guidelines for hypertension diagnosis. The patient needs to be seated some minutes before and during the measurement. The cuff size should be adjusted to the patients' arm circumference and needs to be on the same height level as the patients' sternum during the measurements. Blood pressure is determined to a 2 mmHg accuracy-level. Blood pressure is measured on both arms during the first visit. In both measurements differ more than 10 mmHg, the highest value is taken. After at least 15 seconds, the measurement is repeated during the same visit. The highest mean of the two measurements on the same arm is considered as the actual blood pressure value.
* Patients should fulfil one or more of the following criteria to meet the definition of the metabolic syndrome: 1)Hypertriglyceridemia (serum triglycerides > 1.7 mmol/L); 2) Low High-density lipoprotein (HDL)-cholesterol (serum HDL-cholesterol < 1.04 mmol/L (men) or < 1.29 mmol/L (women)); 3)High fasting glucose (fasting serum glucose > 5.6 mmol/L).
* Patient understands the study procedures, alternative treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion criteria:

* Systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg during one or more screening measurements.
* Body Mass Index (BMI) > 35 kg/m2
* Current smoking or smoking during the previous 3 months
* Use of "recreational" or illicit drugs
* Recent history (within the last year) of alcohol abuse or dependence.
* History of hypersensitivity reactions or intolerance to any (components of) medication used in this trial.
* Current / recent participation (within 30 days of signing informed consent) in a study with an investigational compound or device.
* Laboratory values as follows: Hemoglobin (Hb) < 8,6 mmol/L (men) or < 7.4 mmol/L (women); TSH <0.3 mcIU/mL or > 5.0 mcIU/mL; Potassium < 3,8 mmol/L or > 5,0 mmol/L; Sodium < 136 mmol/L or > 146 mmol/L; MDRD < 60 mL/min/1,73m2
* Medical conditions as follows: Resistant hypertension (blood pressure above target level, despite 3 antihypertensives, including a diuretic); Secondary hypertension; Congestive Heart Failure; Atherosclerotic vascular disease (As per NCEP ATP III and AHA/ACC Guidelines); Cardiac arrhythmia's, for example bradycardia, atrial fibrillation, sick-sinus syndrome, sinoatrial block, atrioventricular block or any other arrhythmia; Obstructive sleep apnea syndrome (OSAS) or a score of 10 or higher on the Epworth Sleepiness Scale questionnaire; Serious liver function disorders (Child-Pugh-Class C); COPD (GOLD classification of severity 2 or higher); Celiac disease or other significant intestinal malabsorption; Malignancy ≤ 5 years prior to signing informed consent, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer; Mental instability or major psychiatric illness; Polyneuropathy or clinical suspicion for autonomic nervous system dysfunction; Any diseases that would limit or complicate study evaluation or participation; Any diseases or screening abnormalities that call for treatment that can not be postponed until after the study period without causing harm.
* Any concomitant medication, particularly antihypertensive co-medication, glucose lowering medication, lipid lowering drugs, systemic corticosteroids, birth control pills and vitamin C or E supplements, but also any other kinds of drugs, including over the counter medication. Exceptions can be made for the following categories of drugs: paracetamol; proton-pump inhibitors; topical creams and unguents that do not lead to uptake of any of the active components into the circulation (in case of steroid creams: class II or lower); inhalation medication, nasal sprays and eye drops that do not lead to uptake of any of the active components into the circulation.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Endothelial function assessed by Flow Mediated Dilation (FMD) | After 8 weeks treatment

SECONDARY OUTCOMES:
Mean 24-hour systolic/diastolic blood pressure Mean day- and night time systolic/diastolic blood pressure | After 8 weeks treatment
Central Blood pressure (estimated with pulse wave analysis) | After 8 weeks treatment
Renin-Angiotensin System (RAS) hormone concentrations | After 8 weeks treatment
Sympathetic nervous system activity, assessed by Muscle Sympathetic Nerve Activity (MSNA) and Heart Rate Variability (HRV) | After 8 weeks treatment
Markers of oxidative stress (concentrations of F2-isoprostanes in urine and oxLDL in plasma) | After 8 weeks treatment
Markers of inflammation (hs-CRP in plasma) | After 8 weeks treatment
Fractional sodium excretion | After 8 weeks treatment
Arterial stiffness (assessed by pulse wave velocity and the pulse wave analysis augmentation index) | After 8 weeks treatment
Adipose tissue function (serum concentrations of adipokines) | After 8 weeks treatment
Lipid metabolism (serum lipid concentrations) | After 8 weeks treatment
Insulin sensitivity, expressed by homeostatic model assessment (HOMA) | After 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: F.L.J. Visseren, Professor (MD PhD), Study Chair — UMC Utrecht; W. Spiering, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Schrover IM, Dorresteijn JAN, Smits JE, Danser AHJ, Visseren FLJ, Spiering W. Identifying treatment response to antihypertensives in patients with obesity-related hypertension. Clin Hypertens. 2017 Oct 24;23:20. doi: 10.1186/s40885-017-0077-x. eCollection 2017. PMID 29085669